CLINICAL TRIAL: NCT00016588
Title: An Open-Label Study to Assess the Anti-HIV-1 Activity of Tenofovir Disoproxil Fumarate (TDF) in Antiretroviral-Naive Patients Who Are Chronically Infected With HIV-1
Brief Title: Tenofovir Disoproxil Fumarate (TDF) in HIV-1 Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 283H; GS-00-917
Record Dates: First submitted 2001-05-17; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-05

CONDITIONS: HIV Infections
Keywords: HIV-1; Adenine; Anti-HIV Agents; Viral Load; Organophosphorus Compounds
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
The purpose of this study is to look at the effectiveness of tenofovir disoproxil fumarate (TDF) in HIV-infected patients who have never taken anti-HIV drugs.

DETAILED DESCRIPTION:
Patients receive TDF.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a plasma viral load (level of HIV in the blood) of 10,000 copies/ml or more.
* Have a CD4 count of 50 cells/mm3 or more.
* Have a negative pregnancy test.
* Agree to use 2 forms of barrier birth control while on the study and for 30 days afterwards.
* Are 18 to 65 years old.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have had treatment with any of the following types of anti-HIV drugs: nucleoside reverse transcriptase inhibitors, nucleotide reverse transcriptase inhibitors (e.g., adefovir dipivoxil or TDF), protease inhibitors, or nonnucleoside reverse transcriptase inhibitors.
* Have received a vaccination within 30 days before study entry.
* Have had a new AIDS-defining illness diagnosed within 30 days before study entry.
* Are taking any of the following: drugs that may cause kidney problems, including aminoglycoside antibiotics, cidofovir, cisplatin, foscarnet, intravenous (IV) amphotericin B, IV vancomycin, oral and IV ganciclovir, and valganciclovir; probenecid; chemotherapy; steroid drugs; interleukin-2; or investigational drugs.
* Are pregnant or breast-feeding.
* Have difficulty taking, absorbing, or tolerating drugs by mouth, as may be shown by long-term nausea or vomiting.
* Abuse alcohol or drugs.
* Have cancer other than Kaposi's sarcoma or basal cell carcinoma.
* Have other infections that need injectable antibiotics within 15 days before study entry.
* Have had kidney or bone disease.
* Have any medical conditions or past treatments that the study investigator believes would make the patient unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York, United States

REFERENCES:
- [Background] Louie M, Hogan C, Hurley A, Captan B, Flaherty J, Lamy P, Balagtas A, Coakley D, Chung C, Ho D. Determining The Relative Efficacy of Tenofovir DF Using Frequent Measurments of HIV-1 RNA During A Short Course of Monotherapy In Antiretroviral Drug Naive Individuals. D, Markowitz M. 9th Conference on Retroviruses and Opportunistic Infections 2002 Feb 24-28